CLINICAL TRIAL: NCT06238037
Title: Bone Mineral Density in Patients With Sarcoidosis
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: SAR4
Record Dates: First submitted 2022-06-03; First posted 2024-02-02 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-12

CONDITIONS: Sarcoidosis; Osteoporosis Risk
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the frequency and risk factors of decreased bone mineral density (BMD) and vertebral fractures in Danish patients with sarcoidosis.

DETAILED DESCRIPTION:
An increased risk of bone fracture has been found in patients with sarcoidosis. Some data showed that the risk of fracture was limited to patients treated with glucocorticoid but data are conflicting and not all studies can prove an increased risk of fracture or bone mineral loss in sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcoidosis
* Signed informed consent

Exclusion Criteria:

* Inability or unwillingness to adhere to the study
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sarcoidosis seen in dep. of Respiratory Diseases and Allergology, Aarhus University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with osteoporosis | At baseline
  Mean BMD at baseline and the distribution of osteopenia osteoporosis and normal scans
Number of patients with osteoporosis | 1 year from diagnosis
  Mean BMD at 1 year and the distribution of osteopenia osteoporosis and normal scans
Number of patients with osteoporosis | 2 years from diagnosis
  Mean BMD at 2 years and the distribution of osteopenia osteoporosis and normal scans
Number of patients with osteopenia | At baseline
  Mean BMD at baseline and the distribution of osteopenia osteoporosis and normal scans
Number of patients with osteopenia | 1 year from diagnosis
  Mean BMD at 1 year and the distribution of osteopenia osteoporosis and normal scans
Number of patients with osteopenia | 2 years from diagnosis
  Mean BMD at 2 years and the distribution of osteopenia osteoporosis and normal scans

SECONDARY OUTCOMES:
Number of participants with vertebral fracture | At baseline
  Proportion of patients with vertebral fracture
Number of participants with vertebral fracture | 1 year from diagnosis
  Proportion of patients with vertebral fracture
Number of participants with vertebral fracture | 2 years from diagnosis
  Proportion of patients with vertebral fracture

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital. Dep. of Respiatory Diseases and Allergology, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No